CLINICAL TRIAL: NCT04355234
Title: Prevalence and Impact of SARS-COV-2 Infection in Pregnant Women, Fetuses and Newborns
Brief Title: Prevalence and Impact of COVID-19 Infection in Pregnant Women, Fetuses and Newborns
Acronym: COVIPREG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: APHP 200448
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2020-04

CONDITIONS: Pregnancy
Keywords: pregnancy; SARS-CoV-2; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, open study with inclusions of 2200 parturients. All parturients divided into 2 groups:
  * 2200 patients whose SARS-Cov-2 status is unknown during pregnancy
  * 300 patients who presented a SARS-CoV-2 infection confirmed by PCR during pregnancy whatever the term
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- all patients (Experimental)
  Interventions: Diagnostic Test: identify SARS-CoV-2 infection by serology
- patients who presented a SARS-CoV-2 infection confirmed by PCR (Experimental)
  Interventions: Biological: collection of biological samples

INTERVENTIONS:
Diagnostic Test: identify SARS-CoV-2 infection by serology — Blood samples at delivery to identify SARS-CoV-2 infection by serology
  Arms: all patients
Biological: collection of biological samples — Creation of a specific collection of biological samples for new investigations thanks to the collection of several biological samples at the time of maternal SARS-CoV-2 infection, at delivery and in the postpartum period in the parturient and her newborn.
  Arms: patients who presented a SARS-CoV-2 infection confirmed by PCR

SUMMARY:
A novel human coronavirus, named SevereAcute Respiratory Syndrome coronavirus 2 (SARS-CoV-2), emerged in China, in late 2019, and is now spreading quickly causing a pandemic. It is usually responsible for a mild infectious syndrome, but patients can also develop pneumonia, acute respiratory failure and other serious complications. To date, very little and controversial literature is available on the impact of SARS-CoV-2 infection on pregnancy, and the potential risk of vertical transmission.

Therefore, the first part of the study, will evaluate the proportion of pregnant woman infected by SARS-CoV-2 during pregnancy over the next six months by performing SARS-CoV-2 serology during pregnancy and at delivery . This information will be correlated to pregnancy and neonatal outcome. The second part of the study 2 will collect sera from several mandatory screening that are kept for one year. Those will be used for assessing the time of the seroconversion and variations of susceptibility to infection with gestational age as well as the impact of social distancing measures.

Concerning neonates born to mothers with documented SARS-CoV-2 infection during pregnancy, only few cases of congenital infections were recently reported because of pneumonia related to SARS-CoV-2 infection and/or positive IgM at birth.

It remains unclear whether neonatal infection can follow transplacental transmission of SARS-CoV-2 during pregnancy and/or through early per- and postnatal exposure, including breast-feeding. In order to investigate these hypotheses, the third part of the study will perform, SARS-CoV-2 PCR tests in a variety of samples collected from infected-mother (symptomatic during the pregnancy and PCR confirmed) and child pairs, at delivery and in the postpartum period.

DETAILED DESCRIPTION:
A novel human coronavirus, named SevereAcute Respiratory Syndrome coronavirus 2 (SARS-CoV-2), emerged in China, in late 2019, and is now spreading quickly causing a pandemic. It is usually responsible for a mild infectious syndrome, but patients can also develop pneumonia, acute respiratory failure and other serious complications. To date, very little and controversial literature is available on the impact of SARS-CoV-2 infection on pregnancy, and the potential risk of vertical transmission. Currently we do not know how many pregnant women may be infected by SARS-CoV-2 and if, as for influenza, they might more likely develop severe infection.

Therefore, the first part of the study, will evaluate the proportion of pregnant woman infected by SARS-CoV-2 during pregnancy over the next six months by performing SARS-CoV-2 serology during pregnancy and at delivery. This information will be correlated to pregnancy and neonatal outcome. The second part of the study 2 will collect sera from several mandatory screening that are kept for one year. Those will be used for assessing the time of the seroconversion and variations of susceptibility to infection with gestational age as well as the impact of social distancing measures.

Concerning neonates born to mothers with documented SARS-CoV-2 infection during pregnancy, only few cases of congenital infections were recently reported because of pneumonia related to SARS-CoV-2 infection and/or positive IgM at birth.

It remains unclear whether neonatal infection can follow transplacental transmission of SARS-CoV-2 during pregnancy and/or through early per- and postnatal exposure, including breast-feeding. In order to investigate these hypotheses, the third part of the study will perform, SARS-CoV-2 PCR tests in a variety of samples collected from infected-mother (symptomatic during the pregnancy and PCR confirmed) and child pairs, at delivery and in the postpartum period.

ELIGIBILITY:
Inclusion Criteria:

* Any pregnant woman giving birth or having a miscarriage after 15 weeks.
* Major patient

Exclusion Criteria:

* Patients not speaking French and not accompanied by a translator
* Patients under curatorship / guardianship
* Refusal to participate in research

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women
Enrollment: 2446 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Seroprevalence or Number of women who are positive for SARS-CoV-2 in parturient woman | at delivery
  Number of women who are positive for SARS-CoV-2

SECONDARY OUTCOMES:
Consequences of SARS-CoV-2 infection in pregnant women and their newborns : Pregnancy outcome, maternal or neonatal complications | 2 months after delivery
  Correlation between exposure to the virus (confirmed by serology) and its impact on pregnancy and its outcome : Pregnancy outcome, maternal or neonatal complications
Assessment of the vertical transmission of SARS-CoV-2 and the possible routes of this transmission in women who are positive for SARS-CoV-2 during pregnancy | at delivery
  Presence of virus (objectified by PCR) in the different biological compartments tested :In the mother: vaginal, anal, amniotic fluid and in the newborn: nasopharyngeal swabs, gastric aspiration, anal swab.
Assessment of the vertical transmission of SARS-CoV-2 and the possible routes of this transmission in women who are positive for SARS-CoV-2 during pregnancy | 5 days after delivery
  Presence of virus (objectified by PCR) in the different biological compartments tested :In the mother: milk and stool samples and in the newborn: nasopharyngeal swabs, urine and stool.
Assessment of susceptibility to infection during the 3 trimesters of pregnancy | 5 days after delivery
  Evaluation of gestational age at SARSCoV-2 infection by performing serology on monthly collected serum samples (samples collected for routine management of pregnancy).
Evaluation of the confinement on the risk of exposure to the virus during pregnancy . | 5 days after delivery
  Study of the methods of confinement by investigation
collection of biological samples for new investigations in women who are positive for SARS-CoV-2 during pregnancy. | 5 days after delivery
  A biobank will be carried out, including the collection of several biological samples at the time of maternal SARS-CoV-2 infection, at delivery and in the postpartum period in the parturient and her newborn
Assessment of the rate of SARS-CoV-2 infection in pregnant women the risk factors for the disease. | at delivery
  Risk factors in uninfected women
Assessment of the rate of SARS-CoV-2 infection in pregnant women the risk factors for the disease. | at delivery
  Risk factors in infected and symptomatic women.
Assessment of the rate of SARS-CoV-2 infection in newborns and the risk factors for the disease. | at delivery
  risk factors in newborns

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Vauloup Fellous, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Tsastaris Vassillis, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vivanti AJ, Couffignal C, Sibiude J, Cordier AG, Tsatsaris V, Rozenberg F, Launay O, Benachi A, De Luca D, Ancel PY, Marcault E, Ville Y, Carrara J, Luton D, Dommergues M, Borie C, Kayem G, Lecomte L, Leruez-Ville M, Perillaud-Dubois C, Biran V, Manchon P, Picone O, Vauloup-Fellous C. Maternal and neonatal outcomes of French prospective multicenter cohort study COVIPREG during the first two COVID-19 waves. J Gynecol Obstet Hum Reprod. 2024 Jun;53(6):102764. doi: 10.1016/j.jogoh.2024.102764. Epub 2024 Mar 16. PMID 38492667
- [Derived] Brebant D, Couffignal C, Manchon P, Duquesne S, Picone O, Vauloup-Fellous C. Transplacental transfer of anti-SARS-CoV-2 neutralizing antibodies in comparison to other pathogens total antibodies. J Clin Virol. 2023 Aug;165:105495. doi: 10.1016/j.jcv.2023.105495. Epub 2023 May 26. PMID 37295035